CLINICAL TRIAL: NCT05933941
Title: Virtual Reality as a Treatment Tool for Chronic Neck Pain in Patients With Fibromyalgia
Acronym: VRTCNPPFM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Principal Investigator, Edurne Úbeda D'Ocasar, Doctor Edurne Úbeda D'Ocasar, Camilo Jose Cela University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CamiloJcURVFM
Record Dates: First submitted 2023-06-19; First posted 2023-07-06 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Fibromyalgia
Keywords: virtual reality; chronic pain; exercises; fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): This group will perform cervical mobility exercises and exercises with virtual reality glasses. 2 sessions will be held per week with a total of 8 sessions
  Interventions: Other: Virtual reality
- Group 2 (Active Comparator): This group will only perform cervical mobility exercises at two sessions per week with a total of 8 sessions.
  Interventions: Other: Exercises
- Control group (No Intervention): This group will not receive any treatment or perform any type of exercise during the duration of this study.

INTERVENTIONS:
Other: Virtual reality — This is a game set in space in which you pilot a spaceship and have to go through rings while dodging meteorites, all controlled by neck movements. Before starting the game, the assigned therapist is in charge of establishing the necessary movement parameters. In addition, the software allows you to modify the difficulty of the game. We will start the first 3 sessions in "easy" mode, where cervical mobility does not exceed 30º. The following 3 sessions will be configured in "medium" mode, reaching 60º of mobility. In the last 2 sessions, we will select the "hard" mode, which not only increases the speed of the spacecraft but also covers the entire range of cervical mobility.
  Arms: Group 1
Other: Exercises — The patients perform mobility and strengthening exercises for the cervical region, in which they are required to complete 1 set of 10 repetitions for each exercise. The patient should rest for at least 30 seconds between exercises.
  Arms: Group 2

SUMMARY:
Fibromyalgia (FM) is a disease characterized by widespread pain, fatigue and cognitive alterations, among other symptoms, neck pain being the most frequent and debilitating. Virtual reality (VR) has emerged as a breakthrough for the treatment of such chronic conditions. The objective of this study is to evaluate the efficacy of VR in the treatment of chronic neck pain in patients with FM. Material and methods: Single-blind randomized clinical trial study. Patients with FM who meet the inclusion criteria will be recruited and will be distributed into three groups (GC, G1, G2). G1 (VR + cervical mobility exercises), G2 (cervical mobility exercises), control group (CG). The treatment will be administered twice a week for 4 weeks. Measurements of variables such as FIQ, EQ-5D, kinesiophobia, pain (VAS and algometer), range of motion (ROM), fatigue and adherence to treatment will be performed.

A follow-up is intended to be carried out 15 days and a month after the end of the study.

DETAILED DESCRIPTION:
RESEARCH QUESTIONS: Can virtual reality combined with exercise improve the quality of life and impact of fibromyalgia? Can exercise performed with VR improve kinesiophobia, cervical range of motion, and pain? Will VR lead to improvements in patients' exercise functional capacity?

The aim is to collect a sample of more than 50 patients with fibromyalgia and cervical pain lasting more than three months. Variables to be collected include cervical range of motion (measured with goniometry), pain (measured with a visual analog scale and pressure algometry at two cervical points), kinesiophobia (TSK questionnaire), impact of fibromyalgia (FIQ), quality of life (EQ-5D), fatigue (BORG visual scale), disability caused by cervical pain (questionnaire), central sensitization (questionnaire), and functional capacity (measured with the "timed-up and go" physical test).

Recruitment was conducted through the Fibromyalgia and Chronic Pain Association of Mostoles. A one-month treatment will be administered with two sessions per week (with at least one day in between), totaling 8 sessions lasting approximately 30 to 40 minutes each. Measurements will be taken before starting the treatment, at the end of the treatment, 15 days after completion, and 30 days after completing the entire treatment.

Subjects will be randomized into three groups: a control group (CG) that will not receive treatment, Group 1 (G1) that will receive cervical mobility exercise combined with exercise using virtual reality (VR), and Group 2 (G2) that will receive cervical mobility exercise alone.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia condition
* present neck pain during the last 3 months

Exclusion Criteria:

* present any pathology that contraindicates the use of virtual reality
* being pregnant at the moment of the study.
* not accepting the informed consent.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) | base line; after finishing the treatment (one month), 15 days after finishing the treatment and 30 days after finishing the treatment.
  visual analogic scale. the maximum value will be 10 and the minimum value will be 0. The higher the score, the more pain the patient will have.
Pain (algometry) | base line; after finishing the treatment (one moth), 15 days after finishing the treatment and 30 days after finishing the treatment.
  Algometer. the maximum value will be 5 and the minimum value will be 0. The higher the score, the less pain the patient will have.
Pain (NDI) | base line; after finishing the treatment (one moth), 15 days after finishing the treatment and 30 days after finishing the treatment.
  Neck Disability Index. Score from 0 to 50. The higher the score, the greater the disability.

SECONDARY OUTCOMES:
Fatigue (BORG) | base line; after finishing the treatment (one month), 15 days after finishing the treatment and 30 days after finishing the treatment.
  Visual Scale BORG. Score from 0 to 10. The higher the score, the greater the perception of fatigue.
Range Of Movement (goniometry) | base line; after finishing the treatment (one moth), 15 days after finishing the treatment and 30 days after finishing the treatment.
  Goniometry of the upper trapezius and suboccipital muscles. Score from 0 to 360º. The higher the degree, the greater the mobility of the patient
Fibromyalgia Impact (FIQ) | base line; after finishing the treatment (one month), 15 days after finishing the treatment and 30 days after finishing the treatment.
  Fibromyalgia Impact Questionnaire. The higher the score obtained, the greater the impact of fibromyalgia on the patient.
Quality of life (EQ-5D) | base line; after finishing the treatment (one month), 15 days after finishing the treatment and 30 days after finishing the treatment.
  EQ-5D Questionnaire. Score from 0 to 15. The higher the score, the worse the quality of life
Central Sensibilization (CSI) | base line; after finishing the treatment (one month), 15 days after finishing the treatment and 30 days after finishing the treatment.
  Central Sensibiliztion Questionnaire. the result obtained ranges from 0 to 100 and the higher the value obtained from the questionnaire the greater the degree of awareness
kinesiophobia (TSK) | base line; after finishing the treatment (one month), 15 days after finishing the treatment and 30 days after finishing the treatment.
  TSK Questionnaire. Each item is scored on a 4-point Likert scale (1 to 4). The response format and numerical values are as follows: (1) strongly agree, (2) disagree, (3) agree, and (4) strongly agree.
  (2) disagree, (3) agree, and (4) strongly agree. The scoring of items 4, 8, 12 and 16 must be inverted to calculate the final score, which can range from 17 to 68.
  17 and 68 and which is obtained by adding the values of the different items.
functional capacity (timed-up and go) | base line; after finishing the treatment (one month), 15 days after finishing the treatment and 30 days after finishing the treatment.
  exercise test (timed-up and go).If the patient takes less than 10 seconds to perform the test, the patient is considered to be at low risk of falling.
  considered low risk of falling. Between 10 and 20 seconds: indicates fragility (risk of falling).
  risk of falling). More than 20 seconds: High risk of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Edurne Ú Úbeda Docasar, Doctor, Principal Investigator — Associate Professor
Locations (1):
- University Camilo José Cela, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No